CLINICAL TRIAL: NCT07051772
Title: Predictive Factors for the Success of Rehabilitation Programs in Chronic Low Back Pain
Acronym: APPROCHE
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2023-1/AD-01
Record Dates: First submitted 2025-03-06; First posted 2025-07-04 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Low Back Pain
Keywords: Biomarkers
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients recruited from Nîmes center
  Interventions: Other: mobility skills testing session

INTERVENTIONS:
Other: mobility skills testing session — A mobility skills testing session using the Qualisys system (Trinoma), when carrying out specific tasks plus 7-day recording of activity using an accelerometer.

SUMMARY:
Chronic low back pain is the leading cause of years lived with disability in the world among 19-49 year olds. The usual progression leads to 15% of acute episodes of persistent pain and more than 50% of persistent activity limitations. Persistent pain lasting between 5 and 7 years causes relatively stable patterns, probably linked to well-known predictive factors of activity limitations such as psychosocial factors (catastrophizing, fears and maladaptive beliefs), physical (deconditioning), professional (fear of returning to work, stress, burden) or personal (financial, insecurity). The effectiveness of treatments is often difficult to predict. Current evidence does not support the use of pharmacological treatments given their low effectiveness and the risks associated with the prescription of non-steroidal anti-inflammatories or opioids, particularly in the chronic phase where the risk of dependence is highest. Thus, international recommendations strongly suggest the use of non-pharmacological therapies, including, physical exercises, rehabilitation, physical and sports activities and spinal manipulations. Most meta-analyses conclude that there is a cumulative effect of the different strategies, without the specific effect of each one being able to be isolated, justifying multidisciplinary protocols. A cornerstone of the management of chronic disabling low back pain therefore relies programs combining physical, cognitive-behavioral, psychological and professional care, most often in dedicated centers. The objective is to empower the patient and promote a change in behavior with regard to the consequences of their pain in the long-term. However, there are very few predictive criteria for the success or failure of these programs, probably because many multiple biological, psychological, and social factors interact over time. Certain models resulting from expert consensus seek to conceptualize these interactions and propose a categorization of these different factors. It is now crucial to validate these categorizations and their relative weight in the progression of patients to best guide their recovery. The aim of this work is to identify the biomarkers predictive of the success of multidisciplinary programs in the short-, medium- and long-term.

ELIGIBILITY:
Inclusion Criteria:

* Patient with chronic low back pain ≥ three months
* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* The patient is participating in a category 1 interventional study, or a study on a medication or medical device without prior approval of the primary investigator
* The patient is in a period of exclusion determined by a previous study
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient followed or treated for a psychiatric, cancerous or orthopedic pathology that risks modifying their course of care
* Pregnant, parturient or breastfeeding patient.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients from the active consultation line in the Physical Medicine and Rehabilitation departments of the University Hospitals of Nîmes, Montpellier and Clermont-Ferrand for chronic low back pain.
Sampling Method: Non-Probability Sample
Enrollment: 333 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Level of disability | Baseline
  Oswestry Disability Index questionnaire. Scoring: 0% to 20%: minimal disability, 20% to 40%: moderate disability, 40% to 60%: severe disability, 60% to 80%: major disability, and 80% to 100 %: bedridden or exaggerated.
Level of disability | Month 6
  Oswestry Disability Index questionnaire. Scoring: 0% to 20%: minimal disability, 20% to 40%: moderate disability, 40% to 60%: severe disability, 60% to 80%: major disability, and 80% to 100 %: bedridden or exaggerated.
Patient age | Baseline
  Years
Patient sex | Baseline
  Male/female
Patient Body Mass Index | Baseline
  Kg/m2
Comorbidities | Baseline
  List of medical pathologies and history of other pathologies of the musculoskeletal system (peripheral osteoarthritis, trauma to the musculoskeletal system, other musculoskeletal disorders).
Pain duration | Baseline
  Months
Professional situation | Baseline
  Description of profession
Work stoppage | Baseline
  Yes/No
Work accident | Baseline
  Yes/No
Disability | Baseline
  Yes/No
Professional Life Satisfaction Scale Socio-economic level | Baseline
Marital status | Baseline
Number of children | Baseline
  Number
Kinesiophobia | Baseline
  Tampa scale
Coping strategies | Baseline
  Coping Strategies Questionnaire
Avoidance Beliefs | Baseline
  Fear-Avoidance Beliefs Questionnaire
Self-efficacy | Baseline
  Pain Self-Efficacy Questionnaire
Catastrophism | Baseline
  Pain Catastrophizing Scale
Acceptance | Baseline
  Acceptance and Action Questionnaire
Anxiety and depression | Baseline
  Hospital Anxiety and Depression Scale
Mobility | Baseline
  Schöber test Finger-to-ground distance
Static endurance of the abdominal muscles | Baseline
  Shirado test, seconds
Isometric endurance of hip and back extensor muscles | Baseline
  Sorensen test, seconds
Central Sensitization | Baseline
  Central Sensitization Inventory
Location of pain | Baseline
  Patient-described using a body diagram
Number and severity of discopathies | Baseline
  Pfirmann classification, measured on MRI
Modic changes on MRI | Baseline
  Present/Absent
Narrow lumbar canal | Baseline
  Yes/No, Measured on MRI
Postural disorder | Baseline
  Yes/No
Scoliosis | Baseline
  Cobb angle
Sagittal balance | Baseline
  Measured using weight-bearing x-rays
Physical Activity | Baseline
  International Physical Activity Questionnaire
Exercise Adherence Rating Scale Sleep | Baseline
  Pittsburgh Questionnaire
Smoking | Baseline
Alcohol consumption | Baseline
Drug use | Baseline
  Yes/No
Knowledge about low back pain | Baseline
  Back Beliefs Questionnaire
Treatment pathway | Baseline
  Description of previous physiotherapy treatments, infiltrations, osteopathy/manual therapy, medicinal treatments

SECONDARY OUTCOMES:
Level of disability | Month 1
  Oswestry Disability Index questionnaire. Scoring: 0% to 20%: minimal disability, 20% to 40%: moderate disability, 40% to 60%: severe disability, 60% to 80%: major disability, and 80% to 100 %: bedridden or exaggerated.
Level of disability | Month 3
  Oswestry Disability Index questionnaire. Scoring: 0% to 20%: minimal disability, 20% to 40%: moderate disability, 40% to 60%: severe disability, 60% to 80%: major disability, and 80% to 100 %: bedridden or exaggerated.
Level of disability | Month 12
  Oswestry Disability Index questionnaire. Scoring: 0% to 20%: minimal disability, 20% to 40%: moderate disability, 40% to 60%: severe disability, 60% to 80%: major disability, and 80% to 100 %: bedridden or exaggerated.
Level of pain | Month 1
  Visual Analog Scale, 0-100
Level of pain | Month 3
  Visual Analog Scale, 0-100
Level of pain | Month 6
  Visual Analog Scale, 0-100
Level of pain | Month 12
  Visual Analog Scale, 0-100
Patient-reported health-related quality of life | Baseline
  Quality of life questionnaire EQ-5D questionnaire, score 0-100
Patient-reported health-related quality of life | Month 1
  EQ-5D questionnaire, score 0-100
Patient-reported health-related quality of life | Month 3
  Quality of life questionnaire EQ-5D questionnaire, score 0-100
Patient-reported health-related quality of life | Month 6
  EQ-5D questionnaire, score 0-100
Patient-reported health-related quality of life | Month 12
  EQ-5D questionnaire, score 0-100
Return to work | Month 12
  Number of days until return to work after end of physiotherapy program
Patients' feelings about symptoms | Month 1
  PGI-C (Patient Global Impression of Change) questionnaire, score 1-7
Patients' feelings about symptoms | Month 3
  PGI-C (Patient Global Impression of Change) questionnaire, score 1-7
Patients' feelings about symptoms | Month 6
  PGI-C (Patient Global Impression of Change) questionnaire, score 1-7
Patients' feelings about symptoms | Month 12
  PGI-C (Patient Global Impression of Change) questionnaire, score 1-7
Mobility abilities of willing patients recruited in the Nîmes center during walking | Baseline
  Three-dimensional optokinetic analysis using Qualisys system
Mobility abilities of willing patients recruited in the Nîmes center during trunk lateral rotations | Baseline
  Three-dimensional optokinetic analysis using Qualisys system
Mobility abilities of willing patients recruited in the Nîmes center during drop jumps | Baseline
  Three-dimensional optokinetic analysis using Qualisys system
Mobility abilities of willing patients recruited in the Nîmes center during Star Excursion Balance Test | Baseline
  Three-dimensional optokinetic analysis using Qualisys system
Mobility abilities of willing patients recruited in the Nîmes center during walking | Month 3
  Three-dimensional optokinetic analysis using Qualisys system
Mobility abilities of willing patients recruited in the Nîmes center during trunk lateral rotations | Month 3
  Three-dimensional optokinetic analysis using Qualisys system
Mobility abilities of willing patients recruited in the Nîmes center during drop jumps | Month 3
  Three-dimensional optokinetic analysis using Qualisys system
Mobility abilities of willing patients recruited in the Nîmes center during Star Excursion Balance Test | Month 3
  Three-dimensional optokinetic analysis using Qualisys system
Moderate-to-vigorous physical activity level of willing patients recruited in the Nîmes center over 7 days | Baseline
  Measured using an accelerometer (ActiGraph, GTX3), minutes
Moderate-to-vigorous physical activity level of willing patients recruited in the Nîmes center over 7 days | Month 3
  Measured using an accelerometer (ActiGraph, GTX3), minutes
Accelerometric parameters of willing patients recruited in the Nîmes center of walking over 7 days | Baseline
  Periods of walking >10 seconds
Accelerometric parameters of willing patients recruited in the Nîmes center of walking over 7 days | Month 3
  Periods of walking >10 seconds
Number of steps of willing patients recruited in the Nîmes center over 7 days | Baseline
  Number, measured using an accelerometer (ActiGraph, GTX3)
Number of steps of willing patients recruited in the Nîmes center over 7 days | Month 3
  Number, measured using an accelerometer (ActiGraph, GTX3)
Duration of a walking period of willing patients recruited in the Nîmes center over 7 days | Baseline
  Minutes, measured using an accelerometer (ActiGraph, GTX3)
Duration of a walking period of willing patients recruited in the Nîmes center over 7 days | Month 3
  Minutes, measured using an accelerometer (ActiGraph, GTX3)
Walking speed of willing patients recruited in the Nîmes center | Baseline
  Km/hour
Walking speed of willing patients recruited in the Nîmes center | Month 3
  Km/hour
Length of strides of willing patients recruited in the Nîmes center | Baseline
  Measured using an accelerometer (ActiGraph, GTX3)
Length of strides of willing patients recruited in the Nîmes center | Month 3
  Measured using an accelerometer (ActiGraph, GTX3)
Duration of strides of willing patients recruited in the Nîmes center | Baseline
  Measured using an accelerometer (ActiGraph, GTX3)
Duration of strides of willing patients recruited in the Nîmes center | Month 3
  Measured using an accelerometer (ActiGraph, GTX3)
Frequency of strides | Baseline
  Medio-lateral and antero-posterior, measured using an accelerometer (ActiGraph, GTX3)
Frequency of strides | Month 3
  Medio-lateral and antero-posterior, measured using an accelerometer (ActiGraph, GTX3)
Acceleration of willing patients recruited in the Nîmes center | Baseline
  Root mean square of the variability of the amplitude of acceleration, measured using an accelerometer (ActiGraph, GTX3)
Acceleration of willing patients recruited in the Nîmes center | Month 3
  Root mean square of the variability of the amplitude of acceleration, measured using an accelerometer (ActiGraph, GTX3)
Gait regularity of willing patients recruited in the Nîmes center | Baseline
  measured using an accelerometer (ActiGraph, GTX3)
Gait regularity of willing patients recruited in the Nîmes center | Month 3
  measured using an accelerometer (ActiGraph, GTX3)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Dupeyron, Principal Investigator — CHU de Nimes
Locations (6):
- France (6):
  - CHU de Clermont Ferrand, Clermont-Ferrand, Auvergne
  - Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard
  - CHU de Montpellier, Montpellier, Occitanie
  - CHU de Nîmes, Nîmes, Occitanie
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Montpellier, Montpellier